CLINICAL TRIAL: NCT00839488
Title: Comparison of Intravenous Pantoprazole and Famotidine for Stress Ulcer Prophylaxis in Patients After Major Abdominal Surgery
Brief Title: Comparison of Intravenous Pantoprazole and Famotidine for Stress Ulcer Prophylaxis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the chief of GS left the hopsital and the successor did't want to keep on this study
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzong-Hsi Lee, Chief of Division of Hepatology and Gastroenterology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FEMH-95-C-011
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Stomach Ulcer
Keywords: pantoprazole; famotidine; stomach ulcer; digestive system surgical procedure
MeSH Terms: conditions — Stomach Ulcer | interventions — Pantoprazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): pantoprazole 40 mg iv qd
  Interventions: Drug: pantoprazole 40 mg iv
- II (Active Comparator): famotidine 20 mg q12h
  Interventions: Drug: famotidine 20 mg iv

INTERVENTIONS:
Drug: pantoprazole 40 mg iv — pnatoprazole 40 mg iv qd
  Other Names: Pantoloc iv
  Arms: I
Drug: famotidine 20 mg iv — famotidine 20 mg q12h
  Other Names: gaster iv
  Arms: II

SUMMARY:
Although stress ulcer is a complication that can cause significant mortality and morbidity in critical patients with risk factors, there is still lack of consensus about its prophylaxis. There are also few data available from Taiwan. H2 blockers are commonly used due to convenience. Some prefer sucralfate (a mucosal protective agent) for the sake of less association with nosocomial pneumonia. Recently, proton pump inhibitors were shown to have good prophylactic effects for stress ulcer. Pantoprazole (iv) is the first intravenous form of proton pump inhibitor that was approved by FDA. There are some reports about its application for treatment of peptic ulcer bleeding. It also has good acid suppression effect in patients under critical care. We expect that intravenous pantoprazole will have a role in stress ulcer prophylaxis.

We will enroll those patients that have received major abdominal surgery and admitted to surgical ICU. After obtaining the consent, we will give them prophylactic drugs for 7 days within 24 hours. They are randomly allocated to 2 groups. Group I: pantoprazole 40 mg iv bolus stat and then qd ; Group II: famotidine 20 mg iv bolus stat and then q12h. We will monitor the following data: operation type & time, APACHE II score, CBC, CXR, stool character and OB test, NG aspirate. If clinical evidence of UGI bleeding occurs, endoscopic examination will be performed. We define the end point as overt bleeding, death or transfer out of ICU. We will compare the prevalence of UGI bleeding and ventilator associated pneumonia in these 2 groups

DETAILED DESCRIPTION:
Patient selection: those receive major abdominal operation (estimated postopeartive ICU stay more than 7 days); agree and give their consent(by their surrogate)within 24 hours after admissionto SICU; those are less than 18 y/o, pregnant, history of allergy to esomeprazole or famotidine, already have GI bleding are excluded Randomized to 2 groups: (1) 1st group to receuve pantoprazole 40 mg iv bolus stat and then qd, (2)2nd group to receive famotidine 20 mg iv bolus stat and then q12h;prophylactically used for 7 days; estimated enrollment of 60 patients for each group Monitoring items: recording opeartion procedure and time; APACHE II score at baseline, CBC、CXR at basleine and qod, stool OB at baseline; NG drainage、sputum、stool character, ICU routine （TPR, BP）;ICU stay，mortality rate at 30 days; EGD perfomed according to decision of attending physician End points: apparant UGI bleeding（tarry stool, meatemesus, large amount(more than 60 ml) of coffee ground from NG、decrease of Hb more than 2g/dl and endoscopically proved lesion）, mortality; ventilator associated pneumonia: new and persistent hazziness in CXR & examination of tracheal aspirate, judged by chest specialist

ELIGIBILITY:
Inclusion Criteria:

* those recieved major abdominal surgery (estimated admission to sirgical ICU more than 7 days); give written consent and was randomized within 24 hours of admission

Exclusion Criteria:

* age less than 18 y/o; pregnant; allergy to famotidine or pantoprazole; have had GI bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
apparant upper gastrointestinal bleeding | 7 days, within the interval of drug prophylaxis

SECONDARY OUTCOMES:
microscopic gastrointestinal bleeding, ventilator associated pneumonia | 7 days, within the interval of drug prophaxis

CONTACTS AND LOCATIONS:
Overall Officials: Tzong Hsi Lee, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Cook DJ, Fuller HD, Guyatt GH, Marshall JC, Leasa D, Hall R, Winton TL, Rutledge F, Todd TJ, Roy P, et al. Risk factors for gastrointestinal bleeding in critically ill patients. Canadian Critical Care Trials Group. N Engl J Med. 1994 Feb 10;330(6):377-81. doi: 10.1056/NEJM199402103300601. PMID 8284001
- [Background] Maier RV, Mitchell D, Gentilello L. Optimal therapy for stress gastritis. Ann Surg. 1994 Sep;220(3):353-60; discussion 360-3. doi: 10.1097/00000658-199409000-00011. PMID 8092901
- [Background] Lu WY, Rhoney DH, Boling WB, Johnson JD, Smith TC. A review of stress ulcer prophylaxis in the neurosurgical intensive care unit. Neurosurgery. 1997 Aug;41(2):416-25; discussion 425-6. doi: 10.1097/00006123-199708000-00017. PMID 9257310
- [Background] Lam NP, Le PD, Crawford SY, Patel S. National survey of stress ulcer prophylaxis. Crit Care Med. 1999 Jan;27(1):98-103. doi: 10.1097/00003246-199901000-00034. PMID 9934901
- [Background] Cook DJ, Reeve BK, Guyatt GH, Heyland DK, Griffith LE, Buckingham L, Tryba M. Stress ulcer prophylaxis in critically ill patients. Resolving discordant meta-analyses. JAMA. 1996 Jan 24-31;275(4):308-14. PMID 8544272
- [Background] Allen ME, Kopp BJ, Erstad BL. Stress ulcer prophylaxis in the postoperative period. Am J Health Syst Pharm. 2004 Mar 15;61(6):588-96. doi: 10.1093/ajhp/61.6.588. PMID 15061430
- [Background] Kantorova I, Svoboda P, Scheer P, Doubek J, Rehorkova D, Bosakova H, Ochmann J. Stress ulcer prophylaxis in critically ill patients: a randomized controlled trial. Hepatogastroenterology. 2004 May-Jun;51(57):757-61. PMID 15143910
- [Background] Tryba M, Cook D. Current guidelines on stress ulcer prophylaxis. Drugs. 1997 Oct;54(4):581-96. doi: 10.2165/00003495-199754040-00005. PMID 9339962
- [Background] Martin LF, Booth FV, Karlstadt RG, Silverstein JH, Jacobs DM, Hampsey J, Bowman SC, D'Ambrosio CA, Rockhold FW. Continuous intravenous cimetidine decreases stress-related upper gastrointestinal hemorrhage without promoting pneumonia. Crit Care Med. 1993 Jan;21(1):19-30. doi: 10.1097/00003246-199301000-00009. PMID 8420726
- [Background] Driks MR, Craven DE, Celli BR, Manning M, Burke RA, Garvin GM, Kunches LM, Farber HW, Wedel SA, McCabe WR. Nosocomial pneumonia in intubated patients given sucralfate as compared with antacids or histamine type 2 blockers. The role of gastric colonization. N Engl J Med. 1987 Nov 26;317(22):1376-82. doi: 10.1056/NEJM198711263172204. PMID 2891032
- [Background] Fabian TC, Boucher BA, Croce MA, Kuhl DA, Janning SW, Coffey BC, Kudsk KA. Pneumonia and stress ulceration in severely injured patients. A prospective evaluation of the effects of stress ulcer prophylaxis. Arch Surg. 1993 Feb;128(2):185-91; discussion 191-2. doi: 10.1001/archsurg.1993.01420140062010. PMID 8431119
- [Background] Pal BK, Roy-Burman P. RNA tumor virus phosphoproteins: subvirion location of the multiple phosphorylated species. Virology. 1977 Dec;83(2):423-7. doi: 10.1016/0042-6822(77)90188-x. No abstract available. PMID 201091
- [Background] Lasky MR, Metzler MH, Phillips JO. A prospective study of omeprazole suspension to prevent clinically significant gastrointestinal bleeding from stress ulcers in mechanically ventilated trauma patients. J Trauma. 1998 Mar;44(3):527-33. doi: 10.1097/00005373-199803000-00020. PMID 9529184
- [Background] Huggins RM, Scates AC, Latour JK. Intravenous proton-pump inhibitors versus H2-antagonists for treatment of GI bleeding. Ann Pharmacother. 2003 Mar;37(3):433-7. doi: 10.1345/aph.1C115. PMID 12639176
- [Background] Hsu PI, Lo GH, Lo CC, Lin CK, Chan HH, Wu CJ, Shie CB, Tsai PM, Wu DC, Wang WM, Lai KH. Intravenous pantoprazole versus ranitidine for prevention of rebleeding after endoscopic hemostasis of bleeding peptic ulcers. World J Gastroenterol. 2004 Dec 15;10(24):3666-9. doi: 10.3748/wjg.v10.i24.3666. PMID 15534928
- [Background] Trepanier EF. Intravenous pantoprazole: a new tool for acutely ill patients who require acid suppression. Can J Gastroenterol. 2000 Nov;14 Suppl D:11D-20D. doi: 10.1155/2000/608413. PMID 11110607